CLINICAL TRIAL: NCT07347587
Title: Study on the Accuracy of Determining the Responsible Vessel in Medium Vessel Occlusive Stroke Based on Multi-type CT Evaluation
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Beijing Hospitals Authority (Unknown)
Responsible Party: Sponsor
Other Study IDs: XMEC-2025-001
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Stroke
Keywords: medium vessel occlusion; Multimodal CT; CTP
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NCCT+CTA group: The attending physicians of neurology (with more than 5 years of experience in neuroimaging interpretation and not relevant to this study), without knowing the final radiological report, DSA, MRI results and clinical manifestations, only used baseline non-contrast CT (NCCT) and CTA to determine whether the included cases had moderate vascular occlusion. And record the qualifying artery
- NCCT+CTA+CTP group: The attending physicians of neurology (with more than 5 years of experience in neuroimaging interpretation and not relevant to this study), without knowing the final radiological report, DSA, MRI results and clinical manifestations, only used baseline non-contrast CT (NCCT) , CTA and CTP to determine whether the included cases had moderate vascular occlusion. And record the qualifying artery

SUMMARY:
To evaluate the accuracy of diagnosing the qualifying artery in patients with medium vessel occlusion stroke based on multimodal CT

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute ischemic stroke, without restrictions on gender
* Age ≥ 18 years old
* The time from onset to treatment is within 24 hours (the onset time is defined as the "last-well-time", and the treatment plan is determined according to the patient's wishes and local clinical experience)
* Before the treatment, CT, CTA and CTP examinations were conducted, and the relevant clinical data were complete.

Exclusion Criteria:

* Patients with acute intracranial hemorrhage
* Patients whose CTP original images cannot be processed by the CTP post-processing software
* Patients for whom the DICOM format image data of CT, CTP original images and MRI images cannot be obtained, or whose image quality is poor due to various reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: According to previous literature reports, the prevalence of MeVO stroke accounts for 18% of ischemic stroke. It is estimated that the sensitivity of NCCT + CTA in diagnosing MeVO is 74%. Based on multimodal CT, the sensitivity for diagnosing moderate vascular occlusive stroke can be increased by 15%, reaching 89%. The test level is bilateral 0.05, and the confidence level 1 - β = 0.8. Then, at least 622 research subjects are required. Among them, the number of patients with MeVO, N1 = 622 * 0.18 = 112 cases.
Sampling Method: Non-Probability Sample
Enrollment: 622 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-03-13 (Estimated); Study Completion 2026-03-13 (Estimated)

PRIMARY OUTCOMES:
The difference in accuracy between the evaluation of MeVO stroke using multimode CT and that using NCCT+CTA | at baseline
  The difference in accuracy between the evaluation of MeVO stroke using multimode CT and that using NCCT+CTA

SECONDARY OUTCOMES:
The time required by the reader to identify the qualifying artery before and after using CTP | at baseline
  The time required by the reader to identify the qualifying artery before and after using CTP
The consistency between the core infarction volume evaluated based on CTP and the final infarction volume obtained from MRI examination within 7 days after the onset | 7 days after the onset
  The consistency between the core infarction volume evaluated based on CTP and the final infarction volume obtained from MRI examination within 7 days after the onset

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No